CLINICAL TRIAL: NCT03470766
Title: Multicentre, Double Blind, Randomised Sham-Controlled Trial of 10kHz High-Frequency Spinal Cord Stimulation for Chronic Neuropathic Low Back Pain (Modulate-LBP)
Brief Title: Sham-Controlled RCT on 10kHz High-Frequency Spinal Cord Stimulation for Chronic Neuropathic Low Back Pain (Modulate-LBP)
Acronym: Modulate-LBP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated early at the request of Sponsors.
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Pain And Neuromodulation Academic Research Centre (PANARC) (Other); University of Exeter (Other); National Institute for Health Research, United Kingdom (Other Government); King's College London (Other); University of Oxford (Other); University of Liverpool (Other); James Cook University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Modulate-LBP
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Chronic Low Back Pain; Neuropathic Pain; Refractory Pain
Keywords: Neuromodulation; HF10; HF-10; Nevro; High-frequency; 10kHz; Spinal Cord Stimulation; CNLBP; Chronic Neuropathic Low Back Pain; Double blind randomised sham-controlled; PANARC; SCS
MeSH Terms: conditions — Neuralgia; Pain, Intractable | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Multicentre, randomised, double-blinded, sham-controlled trial with parallel economic evaluation. Patients will be allocated 1:1 to activated 10kHz SCS plus usual care (intervention) or sham 10kHz SCS plus usual care (control) and followed up to 6 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind. Implanter is blinded, research staff are blinded, subject is blinded. One unblinded research personnel at each recruiting site programming the patients at device activation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Lead (AL) (Active Comparator): One octad lead placed where contacts 4 and 5 span the T9-T10 disc space.
  Interventions: Device: Nevro Senza System (HF10 Therapy)
- Sham Lead (SL) (Sham Comparator): One octad lead implanted subcutaneously behind the IPG and will serve to dissipate the current from the battery
  Interventions: Device: Nevro Senza System (HF10 Therapy)

INTERVENTIONS:
Device: Nevro Senza System (HF10 Therapy) — Nevro 10kHz High Frequency Spinal Cord Stimulation
  Other Names: Neuromodulation; High-frequency stimulation; Nevro; HF-10; HF10; SCS; 10kHz SCS

SUMMARY:
Multicentre, randomised, double-blinded, sham-controlled trial with parallel economic evaluation. Patients will be allocated 1:1 to activated 10kHz SCS plus usual care (intervention) or sham 10kHz SCS plus usual care (control) and followed up to 6 months.

DETAILED DESCRIPTION:
The prevalence of chronic low back pain in the population is estimated to range between at 12% and 28% (1-4). Within this group an estimated 12-15% of adults suffer from chronic neuropathic lower back pain (CNLBP), have relatively greater pain severity, and account for more of the costs of this condition (5,6). This subgroup of people with CNLBP are the focus of the proposed trial.

The National Institute for Health and Care Excellence (NICE) recommends SCS for refractory neuropathic pain (TA159) (7). It is routinely used for people with predominant, neuropathic, radicular pain typically resulting from, or persisting after, spinal surgery (so-called failed back surgery syndrome (FBSS) (8-10). SCS has been shown to be cost effective for this indication (11).

Conventional SCS consists of the insertion of a medical wire (lead) introduced into the epidural space through a needle puncture. The lead is then positioned to target the pain by passing current into the lead from an external power source to generate a pins and needles sensation (paraesthesias) over the painful area. Analgesia occurs when the paraesthesia overlaps and therefore masks the painful area. Once pain reduction is demonstrated, the battery is implanted under the skin of the abdomen, flank or buttock. SCS is most commonly used in the treatment of leg pain of FBSS. However, due to lack of existing evidence and the difficulty of obtaining paraesthesia over the low back, SCS has traditionally not been recommended for treating patients with back pain without previous back surgery (10, 12).

High frequency 10kHz-SCS is a recent major advance in SCS technology. The current is delivered at 10kHz frequency as opposed to the 40 to 60Hz generated by the conventional SCS (13). The key advantages of a higher frequency current are:

10kHz-SCS has been shown to be superior (14) to conventional SCS in targeting residual low back pain following back surgery. Moreover, it does not generate any stimulation related sensations or paraesthesia so is preferred by patients as they are saved from needing to experience these distracting and occasional shocking sensations of conventional SCS. Therefore, 10kHz-SCS allows to smoothly conduct sham controlled or double blind studies in the field of SCS without the need for device modifications.

The lead applicant conducted an uncontrolled, multicentre, single arm study with 83 people with significant low back pain with or without leg pain, implanted with a 10kHz-SCS. At 24 months, the mean reported VAS score for back pain was 3.3 (SD 0.3), compared with 8.4 (SD 0.1) at baseline (pre-implant) and 2.7 (SD 0.3) at 6 months with 60% of subjects reporting >50% back pain relief. Similar improvements were observed in leg pain, disability, sleep and marked reductions in medication intake (15).

In a more recent multicentre RCT, 10kHz-SCS therapy demonstrated superiority to conventional low-frequency SCS in the treatment of post-surgical neuropathic pain. A total of 198 subjects with both back and leg pain were randomised in a 1:1 ratio to a 10 KHz-SCS or conventional SCS. 10kHz-SCS decreased back pain intensity by 67% compared to 44% in the conventional SCS arm (16). This decrease was sustained at 24 months (17).

The above mentioned studies focused on neuropathic back pain in the context of patients with previous spinal surgery. However, a small subset of patients without prior spine surgery that received 10kHz-SCS therapy in both these studies have shown good pain relief and functional improvements in both studies comparable to those with FBSS (14,16).

The investigators hypothesised that patients with CNLBP with no prior spine surgery would benefit from 10kHz-SCS. To evaluate this hypothesis, the investigators initially designed and conducted an open label uncontrolled pilot study in 21 patients with CNLBP and no prior spine surgery. 10kHz-SCS therapy significantly reduced back pain intensity by an average of 5.59 (SD 1.80) (-72.6% vs baseline) at 12 months in medically refractory low back pain patients with no past history of spine surgery. 90% of the implanted patients were classified as responders (i.e. VAS back pain reduction >50%) at 12 months. The investigators also observed a significant increase in physical function scores and health-related quality of life at one year post 10kHz-SCS implant. Mean pain intensity was reduced by 73% and disability measured by the Oswestry Disability Index was reduced by 48%. Opioid medication intake decreased by 64% and mean EQ-5D quality of life scores improved from 0.16 to 0.47. More importantly 75% of patients were able to return to employment(18). This improvement was sustained at 3 years follow up (19).

Following these promising results, the investigators now intend to undertake a fully powered RCT to confirm our hypothesis that 10kHz-SCS is beneficial for CNLBP patients with no prior back surgery.

To date 10kHz-SCS has not been formally tested against a sham control condition in order to isolate the therapeutic effects from those induced by placebo. It is very possible that some of the benefit reported may be due to a placebo effect (enhanced by a surgical procedure) or reporting bias in either the patient or assessor. The investigators have therefore specifically designed this fully powered double blind randomised sham controlled trial of 10kHz-SCS to address this major methodological limitation of previous studies.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over the age of 18
2. Onset of low back pain > 12 months
3. Low back pain intensity > 60 out of 100mm on pain visual analogue scale (VAS)
4. Presence of clear component of neuropathic pain based on a PainDETECT Questionnaire score of >19 (we will monitor this inclusion criteria in the early stage of the trial and revise if necessary)
5. Degenerative disc disease confirmed by imaging or internal disc disruption as confirmed by discography
6. On stable pain medications, as determined by the Investigator, for at least 28 days prior to enrolling in this study and not change medication dosage without consulting Investigator
7. Legally able to provide informed consent
8. Able to comply with study-related requirements, procedures and visits

Exclusion Criteria:

1. Had previous spinal surgery
2. Chronic widespread pain
3. Subject has an active implanted device, whether turned on or off (e.g. pacemaker, intrathecal pump, deep brain stimulator etc.)
4. A current diagnosis of a progressive neurological disease such as multiple sclerosis, chronic inflammatory demyelinating polyneuropathy, rapidly progressive arachnoiditis, rapidly progressive diabetic peripheral neuropathy, brain or spinal cord tumour, or severe/critical central or foraminal spinal stenosis
5. Mechanical spine instability detected by a clinician (validation by flexion/extension films of lumbar spine within the past 6 months showing 4 mm or more translational movement or excessive angular movement manifested by >5 degrees segmental angular movement) e.g. any forms of spondylolisthesis
6. A medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints, as determined by the Investigator
7. Bleeding diathesis such as coagulopathy or thrombocytopenia
8. Immunocompromised and at an increased risk for infection
9. Systemic infection or local infection that would contraindicate SCS placement
10. Metastatic malignant disease or active local malignant disease
11. Pregnant (if female and sexually active, subject must be using a reliable form of contraception, be surgically sterile or be at least 2 years post-menopausal)
12. Active alcohol, marijuana, recreational or prescription drug abuse or dependence or unwilling to stop/reduce excessive inappropriate medication.
13. Evidence of an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance of intervention and/or ability to evaluate treatment outcome as determined by the Investigator
14. Concomitant participation in another clinical trial (surgery, device or drug)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Mean VAS Back Pain (7 Day Subject VAS Pain Diary) | 6 months post randomisation
  Changes in mean VAS back pain between intervention and control at 6 months post-randomisation

SECONDARY OUTCOMES:
Oswestry disability index (v2.1a) | 1, 3, and 6 months post randomisation
  To compare disability between intervention and control at 1, 3, and 6 months post-randomisation.
PHQ-9 Questionnaire | 1, 3, and 6 months post randomisation
  To compare depression between intervention and control at 1, 3, and 6 months post-randomisation.
PSQI Questionnaire | 1, 3, and 6 months post randomisation
  To compare sleep quality between intervention and control at 1, 3, and 6 months post-randomisation.
PGIC Questionnaire | 1, 3, and 6 months post randomisation
  To compare patients' global impression of change between intervention and control at 1, 3, and 6 months post-randomisation.
EQ-5D Questionnaire | 1, 3, and 6 months post randomisation
  To compare health-related quality of life between intervention and control at 1, 3, and 6 months post-randomisation.
Medication Usage | 1, 3, and 6 months post randomisation
  To compare medication usage between intervention and control at 1, 3, and 6 months post-randomisation.
Sensation Map | 1, 3, and 6 months post randomisation
  To compare sensation maps between intervention and control at 1, 3, and 6 months post-randomisation.
Healthcare utilisation, work status, work absence, and out of pocket expenses | 6 months post randomisation
  To compare the cost-effectiveness of 10kHz-SCS between intervention and control at six months post-randomisation.
Safety/Adverse Events | 6 months post randomisation
  To compare complications and adverse events at 6-months post-randomisation between intervention and control.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Guy's and St Thomas Hospital, London
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473
- [Derived] Al-Kaisy A, Royds J, Palmisani S, Pang D, Wesley S, Taylor RS, Cook A, Eldabe S, McCracken L, Duarte R, Fairbank J. Multicentre, double-blind, randomised, sham-controlled trial of 10 khz high-frequency spinal cord stimulation for chronic neuropathic low back pain (MODULATE-LBP): a trial protocol. Trials. 2020 Jan 28;21(1):111. doi: 10.1186/s13063-019-3831-4. PMID 31992344